CLINICAL TRIAL: NCT01185899
Title: The Usefulness of High-frequency QRS Analysis in the Evaluation of Patients Presenting to the Emergency Department With Chest Pain
Brief Title: Usefulness of High-frequency QRS Analysis in the Evaluation of Patients With Chest Pain
Status: Completed | Type: Observational
Sponsor: Ori Galante (Other)
Collaborators: BSP Biological Signal Processing Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Ori Galante, Co-PI, Soroka University Medical Center
Organization: Soroka University Medical Center (Other)
Other Study IDs: sor505310ctil
Record Dates: First submitted 2010-08-18; First posted 2010-08-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Acute Coronary Syndrome; STEMI; NSTEMI; Unstable Angina; Chest Pain
Keywords: heart attack; acute myocardial infarction; STEMI; NSTEMI; Unstable Angina; suspected acute coronary syndrome; Non-ischemic chest pain
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Angina, Unstable; Chest Pain; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected ACS patients: Patients presenting with chest pain to the Emergency Department, who are suspected of having ACS, will be asked to participate in the study.

SUMMARY:
Accurate detection of a heart attack (an acute myocardial infarction) is one of the most pressing needs in medicine. Recordings of the electrocardiogram (ECG) (electrical activity of the heart) are one of the first tools used to diagnose a heart attack, but the ECG is not very accurate, especially at the beginning of a heart attack. A new technique for analysing a special part of the ECG may provide more accurate detection of a heart attack. The study hypothesis is that this new technique, the HFQRS analysis, will provide important additional information to that available from the regular ECG.

DETAILED DESCRIPTION:
Chest pain is one of the leading reasons for hospital emergency department (ED) visits worldwide. In the United States (US), over 6 million people annually undergo evaluation in the ED for acute chest pain. Despite the wealth of knowledge available about acute coronary syndrome (ACS), this condition continues to be among the most difficult to predict or diagnose. Nearly half of patients hospitalized for unstable angina eventually receive a non-cardiac-related diagnosis. Nonetheless, 2-8% of patients with myocardial infarction (MI) are inappropriately discharged from the ED and mortality rates among patients with an MI who were mistakenly sent home are disproportionately higher (25-33%) than those among patients who were admitted.

Although the ECG is a mainstay in the management of suspected ACS, it has major limitations in both sensitivity and specificity for diagnosis of ACS. The initial 12-lead ECG in the ED is often non-diagnostic in ACS patients, especially in non-ST elevation MI (NSTEMI) and unstable angina (UA), and therefore cannot rule-out ischemia or infarction. Elevation in serum biomarkers is usually not detectable for 4-6 hours after an MI, and some patients do not show a biomarker elevation for as long as 12 hours. Consequently, new clinical tools for early risk stratification of patients with acute chest pain are being sought.

Conventional analysis of ST segment deviations aims to detect repolarization abnormalities. However, ischemia may also bring about changes in the depolarization phase of the electrical cardiac cycle. These depolarization changes can be detected and quantified using analysis of the high-frequency components of the QRS complex (HFQRS). HFQRS analysis has been previously reported to be a sensitive method for detection of demand ischemia during exercise testing. Preliminary studies have shown that HFQRS-derived indices can also identify supply ischemia caused by prolonged balloon occlusion, and transient ischemic episodes in patients with chest pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chest pain, suspected to have ACS
* Duration of chest pain greater than 20 minutes
* Time from onset of chest pain less than 12h
* Signed an informed consent

Exclusion Criteria:

* History of trauma or any other evident medical cause of chest pain
* Prior coronary artery bypass graft
* Pre-excitation syndrome (example WPW)
* Atrial Fibrillation or significant ventricular arrhythmia
* Bundle branch block, intraventricular conduction delay or
* QRS duration greater than 120 ms
* Implanted pacemaker or defibrillator
* Patients who received fibrinolytic therapy, glycoprotein IIb or IIIa inhibitors before the initial ECG recording

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients arriving to the emergency department of Soroka University Medical Center with chest pain that is suspected of being due to acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2010-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
diagnosis or rule-out of acute coronary syndrome | diagnosis or rule-out of ACS will be determined at two time points: 1) upon diacharge when discharge diagnosis is determined. Follow up information will be obtained one month post discharge
  The primary end-point of the study is definite discharge diagnosis or rule-out of acute coronary syndrome, based on cardiac biomarkers, ECG changes, clinical symptoms and cardiac imaging tests.

CONTACTS AND LOCATIONS:
Overall Officials: Doron Zahger, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

REFERENCES:
- [Derived] Galante O, Amit G, Granot Y, Davrath LR, Abboud S, Zahger D. High-frequency QRS analysis in the evaluation of chest pain in the emergency department. J Electrocardiol. 2017 Jul-Aug;50(4):457-465. doi: 10.1016/j.jelectrocard.2017.02.009. Epub 2017 Feb 20. PMID 28341306